CLINICAL TRIAL: NCT02811991
Title: A PhaseⅡ/ Ⅲ Seamless Study to Evaluate Efficacy and Safety of Paracetamol Injection as Adjuvant to Morphine-based Postoperative Analgesia-Multicentered, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: A PhaseⅡ/ Ⅲ Seamless Study to Evaluate Efficacy and Safety of Paracetamol Injection as Adjuvant to Morphine-based Postoperative Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-DYXAJF-Ⅲ
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Post-operative Analgesia
Keywords: paracetamol; post-operative analgesia
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental:Paracetamol Injection (Active Comparator): 325mg(32.5mL)or 500mg(50mL) iv q6h according to assignment
  Interventions: Drug: Paracetamol injection; Drug: Morhpine PCA
- Placebo:Normal Saline Injcetion (Placebo Comparator): 32.5mLor 50mL iv q6h according to assignment.
  Interventions: Drug: Normal Saline injection; Drug: Morhpine PCA

INTERVENTIONS:
Drug: Paracetamol injection — 325mg(32.5mL) or 500mg(50mL) iv q6h,4 doses in 24h.Infushion time≥15min.
  Arms: Experimental:Paracetamol Injection
Drug: Normal Saline injection — 32.5mL or 50mL iv q6h,4 doses in 24h.Infushion time≥15min.
  Arms: Placebo:Normal Saline Injcetion
Drug: Morhpine PCA — Morphine PCA will be connected upon the first dose of study drug(roughly 30min prior to the completion of would suture). Morphine PCA is set as follows:1mg bolus every 5min with background infusion of 0.25mg/h and maximal dose<25mg/4h.

SUMMARY:
Paracetamol,a classical analgesic agent,constitutes an essential component of multi-modal analgesia. This medication is generally safe, well tolerated and effective within recommended daily dose.The purpose of the study is to evaluate the efficacy and safety of Paracetamol Injection as adjuvant to morphine-based post-operative analgesia, as well as to explore the reasonable dosage of paracetamol among Chinese population under above-mentioned circumstance.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 70 years inclusively, male or female;
* Patients scheduled for open abdominal surgery(such as gall bladder, lower abdominal investigative surgery), gynecologic surgery(such as trans-abdominal hysterectomy), orthopedic surgery(such as replacement and reconstruction of knee, hip or shoulder joint), with anticipated need for post-operative iv. morphine analgesia≥24h;
* 18kg/m2≤BMI≤30 kg/m2;
* Classified as ASA risk class I, II according to the American Society of Anesthesiologists;
* Able to understand the study procedures and the use of the pain scales, able to operate a patient controlled analgesia (PCA) device and to communicate meaningfully with the study observer and staff;
* Patients free of any contraindication to the study drugs, morphine and to the standardized anesthesia protocol;
* Clearly understand the procedure of study, voluntarily participate and provided written consent form.

Exclusion Criteria:

* Impaired liver function (ALT and/or AST > 2 x upper limit of normal range, or TBIL≥1.5 x upper limit of normal range);
* Impaired renal function(Serum Creatinine >176μmoL/L), or undergoing dialysis within 28 days before surgery;
* Patients at high risk for bleeding, including congenital hemorrhagic disease(such as Hemophilia), Thrombocytopenia(CBC PLT<30×109/L), Qualitative Plateletdefects(such as ITP, DIC, congenital abonormal platelet), or clinically significant active bleeding;
* Abnormal resting ECG, judged as not eligible for entry by investigator;
* Hypertensive patients not achieving satisfactory BP control under hypertensive medication(Sitting SBP≥160mm Hg, and/or DBP≥105mm Hg during screen period);
* Sitting SBP≤90mm Hg during screening period;
* Diabetic Patients not achieving satisfactory blood glucose control(FBG≥11.1moL/L during screening period);
* Known history of bronchial asthma, pulmonary heart disease or heart failure;
* Participation in other trials within 30 days;
* Pregnant women or women in lactation;
* Patients not eligible due to other reasons judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09-14 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Total morphine use in 24 hours | 24h after the 1st dose of study drug
  Total morhpine use(including PCA and emergency morphine use)in 24 hours.

SECONDARY OUTCOMES:
Pain Intensity VAS AUC(0-24h) at rest | 0-24h PI VAS AUC(mesured at 1h、3h、6h、12h、24h after the 1st dose of study drug)
Pain Intensity VAS AUC(0-24h) at movement | 0-24h PI VAS AUC(mesured at 1h、3h、6h、12h、24h after the 1st dose of study drug)
Incidence of mophine-related ADR | 0-24h after the 1st dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Fei Liu, Ph.D, Principal Investigator — West China Hospital
Locations (16):
- China (16):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The South West Hospital, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Millitary Command, Fuzhou, Fujian
  - Liuzhou General Hospital, Liuchow, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - the Third Xiangya Hospital of Central South University, Changsha, Hunan
  - No.1 People's Hospital of Chenzhou City, Chenzhou, Hunan
  - Affiliated Hospital,Jiangnan University, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tongji Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Ningbo No.2 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yin F, Ma W, Liu Q, Xiong LL, Wang TH, Li Q, Liu F. Efficacy and safety of intravenous acetaminophen (2 g/day) for reducing opioid consumption in Chinese adults after elective orthopedic surgery: A multicenter randomized controlled trial. Front Pharmacol. 2022 Jul 22;13:909572. doi: 10.3389/fphar.2022.909572. eCollection 2022. PMID 35935863